CLINICAL TRIAL: NCT00299091
Title: Open, Parallel and Randomised Pilot Clinical Trial to Evaluate the Utility of the Therapeutic Monitoring of Plasma Levels of Efavirenz in Hiv-Infected Patients Initiating an Antiretroviral Treatment Regimen With Sustiva
Brief Title: Modification of Doses of Efavirenz According to Its Blood Concentration in HIV Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Dr . BONAVENTURA CLOTET, Dr. Bonaventura Clotet, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: startTDM-EFV; 2005-002493-30
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: HIV
Keywords: Therapeutic drug monitoring; Treatment Naive; Treatment Experienced; HIV
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Efavirenz capsules 600 mg
- Experimental (Experimental): Modification of doses of efavirenz guided by its plasma concentration (therapeutic drug monitoring)
  Interventions: Drug: Efavirenz capsules 200 mg and 600 mg

INTERVENTIONS:
Drug: Efavirenz capsules 200 mg and 600 mg — Modification of doses of efavirenz guided by its plasma concentration (therapeutic drug monitoring)
  Other Names: Sustiva
  Arms: Experimental

SUMMARY:
This is a study on the utility of the modification of doses of efavirenz guided by its plasma concentration (therapeutic drug monitoring) in HIV-infected patients initiating treatment with Sustiva.

DETAILED DESCRIPTION:
Currently, efavirenz is dosed systematically, without taking into account the individual characteristics of each individual patient. However, plasma concentration of efavirenz may widely vary between different subjects that receive the same dose of the drug (interindividual variability).

Therapeutic drug monitoring (TDM) signifies individualised pharmacological dosing, based on the plasma levels that each patient presents. This strategy has been broadly used in the field of the treatment of other medical conditions and is acquiring growing interest in the field of antiretroviral treatment. Thus, the use of TDM for the treatment of naïve patients with nelfinavir or with indinavir has translated into an increase in the proportion of individuals with suppressed viral load and also into a reduction in HAART-induced adverse events . However, data on the utility of the therapeutic monitoring of the levels of efavirenz in HIV-infected patients are very scant.

On the basis of the above, it might be thought that the modification of the doses of efavirenz, guided by its plasma concentration, in patients receiving this drug and whose plasma levels of efavirenz are outside the therapeutic range, might improve the tolerability of the treatment without compromising virological efficacy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 patients.
* According to the criteria of the treating physician, the need to initiate a regimen of antiretroviral treatment that includes efavirenz (both antiretroviral-naive patients and others on treatment with protease inhibitors switching to efavirenz for salvage reasons or for simplification of the anti-retroviral therapy are included).
* Absence of opportunistic infections and/or tumours in the three months prior to inclusion.

Exclusion Criteria:

* History of allergic hypersensitivity to the investigational drug.
* History of previous failure with antiretroviral treatment with non-nucleoside reverse transcriptase inhibitors or previously documented resistance to efavirenz
* History of psychiatric comorbidity which, in the investigator's opinion, renders the use of efavirenz inadvisable.
* Active consumption of alcohol (>50 g/day) or other illegal drugs (except cannabis)
* Suspicion of unsuitable compliance with the antiretroviral treatment.
* Pregnant women or breast-feeding mothers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who need to interrupt treatment with efavirenz due to virological failure | after 96 weeks of follow-up

SECONDARY OUTCOMES:
The proportion of patients who need to interrupt treatment with efavirenz due to adverse side effects | after 96 weeks of follow-up
To determine the incidence of adverse events and the toxicity profile (haemogram, AST/ALT/FA/GGT, creatinine, urea) | during the 96 weeks of follow-up
To evaluate the proportion of patients with plasma levels of efavirenz between 1.0 and 4.0 mg/L | during the 96 weeks of follow-up
To evaluate the relationship between the appearance of secondary events during treatment with efavirenz and the patients' demographic and clinical characteristics, as well the plasma concentration of efavirenz | during the 96 weeks of follow-up
To evaluate the variations in CD4 and CD8 lymphocyte count | during the 96 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD, PhD, Principal Investigator — Lluita Sida Foundation-HIV Unit
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain